CLINICAL TRIAL: NCT01125436
Title: A Randomized Placebo Controlled Trial of Vitamin D Therapy in Patients With Heart Failure
Brief Title: A Trial of Vitamin D Therapy in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1KL2RR024990 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Aerobic Capacity; Strength
MeSH Terms: conditions — Heart Failure | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Experimental): Nutritional supplement
  Interventions: Dietary Supplement: Cholecalciferol
- placebo (Placebo Comparator): Weekly placebo plus 800 calcium daily
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 50,000 units of oral vitamin D3(cholecalciferol) weekly plus 800 calcium daily
  Other Names: Vitamin D
  Arms: Cholecalciferol
Dietary Supplement: Cholecalciferol — Weekly placebo plus 800 calcium alone
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if vitamin D will improve physical performance in older adults with heart failure.

DETAILED DESCRIPTION:
The study is designed as a short pilot study which will assess safety and efficacy of high dose Vitamin D therapy in a heart failure population.

A 6 month randomized double blind placebo-controlled trial of 50,000 units of oral vitamin D3(cholecalciferol) weekly plus 800 calcium daily vs. weekly placebo plus 800 calcium alone in 64 heart failure (HF) patients > 50 years old. This design was chosen over a cross-over design due to the long wash-out period for vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) class II-IV
* Able to walk
* Serum 25OHD level 37.5 ng/ml or less
* Fully titrated on heart failure medications

Exclusion Criteria:

* Osteoporosis
* Primary hyperparathyroidism or hypercalcemia.
* Nephrolithiasis
* Hemo or peritoneal dialysis and/or creatinine of > 2.5
* Current use of daily vitamin D greater than 400 IU, corticosteroids, parathyroid hormone (PTH), androgen or estrogen
* Current illicit drug user or > 3 alcoholic drinks a day
* Metastatic or advanced cancer
* Myocardial infarction in the preceding 6 months
* Medications which can lower vitamin D levels or bioavailability

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Boxer, MD, Principal Investigator — Case Western Reserve Univerity
Locations (1):
- University Hospitals/Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment May 2007-April 2011 outpatient heart failure and cardiology clinics
Groups:
- Cholecalciferol + Calcium: Nutritional supplement
  Cholecalciferol : 50,000 IU weekly for 6 months
- Placebo +Calcium: Cholecalciferol : Placebo weekly for 6 months
Period: Overall Study
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Started | 31 | 33
Completed | 19 | 21
Not Completed | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Cholecalciferol + Calcium: Participants received vitamin D
- Placebo + Calcium: Participants received placebo
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol + Calcium | Placebo + Calcium | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10.6) | 66.0 (10.4) | 65.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Peak VO2
Description: Cardiopulmonary stress testing with the Peak VO2 representing maximal aerobic capacity
Time Frame: change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Number analyzed (Participants) | 24 | 23
ml/kg/min | -.17 (2.07) | -.68 (1.85)

2. Secondary Outcome: Leg Proximal Muscle Strength
Description: Strength of the proximal lower extremity muscles measured by peak torque Nm/kg adjusted for body weight in flexion and extension
Time Frame: change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: newton-meters/kg
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Number analyzed (Participants) | 24 | 24
newton-meters/kg
  Flexion 60°s-1 | 1.6 (17.2) | 5.1 (8.8)
  Extension 60°s-1 | 5.2 (29.7) | 3.5 (17.1)

3. Secondary Outcome: 6 Minute Walk Distance
Description: The six-minute walk test is a reliable and valid test of aerobic capacity, predictive of morbidity and mortality outcome, and correlates with Activity of Daily Living (ADL) and Quality of Living (QOL).
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Number analyzed (Participants) | 24 | 26
meters | 59 (282) | 36 (228)

4. Secondary Outcome: Timed Get Up and Go
Description: stand from chair walk 3 meters, return to chair and sit
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Number analyzed (Participants) | 25 | 25
seconds | -0.2 (3.3) | -1.0 (3.3)

5. Other Pre Specified Outcome: Serum Aldosterone
Description: Serum for aldosterone will be drawn at baseline, 3, and 6 months, and processed according to lab protocol.
Time Frame: change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Number analyzed (Participants) | 31 | 31
ng/dl | 3.7 (13.65) | -0.1 (15.55)

6. Other Pre Specified Outcome: Plasma Renin Activity
Description: Serum for renin will be drawn at baseline, 3, and 6 months, and processed according to lab protocol.
Time Frame: change in renin from baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/ml/hr
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Number analyzed (Participants) | 29 | 28
ng/ml/hr | 1.3 (13.84) | -2.5 (15.25)

ADVERSE EVENTS:
Arm/Group | Cholecalciferol + Calcium | Placebo +Calcium
Serious Adverse Events (participants affected / at risk) | 3/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol + Calcium (N=31) | Placebo +Calcium (N=33)
hospitalization (Cardiac disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No